CLINICAL TRIAL: NCT00341471
Title: Adolescent Pregnancy Prevention: Building Futures for Youth
Brief Title: Building Futures for Youth - Phase III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906078; 06-CH-N078
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-18

CONDITIONS: Adolescent Pregnancy
Keywords: School; Sixth Grade; Curricular; Howard University; D.C.; Adolescent Pregnancy; Intervention

INTERVENTIONS:
Procedure: Risk Behavior Prevention Intervention Program

SUMMARY:
The Building Futures for Youth (BFY) project is a pilot intervention program for 6th grade students and their parents in the District of Columbia public school system. The full intervention will include students in the 6th, 7th and 8th grades. The primary overall goal of the project is to help students learn to make healthy life choices and delay sexual initiation.

Sixth-grade children and parents in four Washington, D.C., public schools will be recruited for this study. Children from two schools will participate in the BFY intervention program and children from two other schools will serve as controls. Participants are guided through three study phases, with each phase spanning one school year, as follows:

Sixth-grade students are given a foundation in goal setting, decision-making and communication skills. They gain knowledge about puberty, reproduction, and the negative consequences associated with having a child at a young age. They learn strategies for getting out of situations in which they feel pressured to engage in sexual activity. Through lessons, activities, and discussions they are given tools to answer the following questions:

* Who am I? Students engage in self-reflection activities and discussions that allow them to become aware of their values, beliefs and strengths, increasing self-esteem and a positive self-image.
* What do I want for my life? Students engage in goal-setting activities, creating short-term and long-term goals and mapping out the necessary steps to achieve the goals.
* How do I get there? Students are instructed in decision-making, problem-solving and communication skills.
* How can having sex too early affect my life and the goals I want to achieve? Students explore the negative impact that engaging in sexual activity too early and getting pregnant or getting someone pregnant can have on their emotional, social and financial lives.

Seventh grade students are given the tools and skills necessary to deal with a variety of challenges they may experience during their developmental years. They receive comprehensive sex education, in conjunction with life skills such as relationship negotiation, dating skills, violence prevention and problem-solving skills.

Eighth grade students are guided through a series of activities that encourage students to translate knowledge gained in the 6th and 7th grade phases into long-term behavioral changes and risk reduction. Activities include writing and performing skills, creating an informational pamphlet, designing T-shirts and creating poetry that affirms the BFY message.

In addition, students participate in a program of community service projects, such as the Anacostia River clean-up coordinated by the Earth Conservation Corps and Martin Luther King Day events coordinated by Howard University's Community Association and Project Change.

Parents are provided skills training and information on a variety of issues relating to adolescent sexuality, parental monitoring and parent-child communication.

DETAILED DESCRIPTION:
The Adolescent Pregnancy Prevention Project, or Building Futures for Youth, is embarking on a pilot year in order to test the effectiveness of a revised children's intervention for Grade 6. Although there was some evidence of a positive effect of the intervention for girls during Phase II, there were no significant effects for boys. In light of these findings, BFY will spend the current project year piloting a revised classroom intervention as well as a newly adapted after-school intervention component.

ELIGIBILITY:
* INCLUSION CRITERIA:

The target population for the pilot year is primarily African-American children who are sixth grade students at the participating schools.

Active parental consent will be required for all participants and will be required for all participants and will be required separately for participation in the classroom intervention session and participation in Club SERVE.

All children who can understand English will be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2006-01-18; Primary Completion 2008-10-08 (Actual); Study Completion 2008-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Howard University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Koo HP, Rose A, El-Khorazaty MN, Yao Q, Jenkins RR, Anderson KM, Davis M, Walker LR. Evaluation of a randomized intervention to delay sexual initiation among fifth-graders followed through the sixth grade. Sex Educ. 2011 Feb;11(1):27-46. doi: 10.1080/14681811.2011.538146. PMID 21857793